CLINICAL TRIAL: NCT02957747
Title: Addressing the Health Concerns of VA Women With Sexual Trauma
Acronym: SHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VISN 17 Center of Excellence (U.S. Federal Agency)
Collaborators: Brown University (Other); Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Suzannah Creech, Psychologist, VISN 17 Center of Excellence
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00614
Record Dates: First submitted 2016-09-21; First posted 2016-11-08 (Estimated); Results first posted 2020-01-02 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Stress Disorders, Post-Traumatic; Intimate Partner Violence; Alcohol-Related Disorders
Keywords: Women Veterans; Sexual Trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcohol-Related Disorders; Sexual Trauma | interventions — Safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safety and Health Experiences Program (Experimental): Participants in the SHE arm of the study will receive a web-based intervention utilizing motivational interviewing and education.
  Interventions: Behavioral: SHE
- Control (No Intervention): Participants randomized to this arm will receive referrals to VA and community resources

INTERVENTIONS:
Behavioral: SHE — SHE is a computer-delivered intervention (Safety and Health Experiences Program; SHE) that will provide a screening and brief behavior intervention for women Veterans with any lifetime ST. More specifically, the intervention, SHE, will address interrelated health concerns for women Veterans with ST (i.e. alcohol misuse, IPV, and PTSD). SHE will provide individualized assessment, feedback, and referrals for women Veterans with any lifetime ST. SHE will take place within a primary care setting.
  Other Names: Safety and Health Experiences program
  Arms: Safety and Health Experiences Program

SUMMARY:
Lifetime sexual trauma (ST) (i.e., behaviors that range from unwanted sexual touching to attempted or completed rape) is a significant social and public health problem among women Veterans. For women Veterans, lifetime ST can occur prior to, during or after military service. ST is associated with multiple difficulties and risks, including posttraumatic stress disorder (PTSD), intimate partner violence (IPV), and alcohol misuse. Providing an effective, integrated, and low-cost intervention that targets ST-related risks for women Veterans with lifetime ST would advance clinical care for these vulnerable women.

This research will develop and assess a computer-delivered intervention (Safety and Health Experiences Program; SHE) that will provide a screening and brief behavior intervention for women Veterans with any lifetime ST. More specifically, the intervention, SHE, will address interrelated health concerns for women Veterans with ST (i.e. alcohol misuse, IPV, and PTSD). SHE will be designed to provide individualized assessment, feedback, and referrals for women Veterans with any lifetime ST. SHE will take place within a primary care setting. Primary care visits are frequent points of health care contact for women Veterans making the visit itself the ideal, and possibly only, opportunity to provide behavioral interventions.

This study will lay the groundwork for a larger clinical trial of the SHE program in multiple VA primary care settings. If effective, the intervention, SHE, represents an innovative and low cost service for early identification and intervention that could be implemented nationwide with ease and speed to address the needs of women Veterans with lifetime ST. The long-term goal of the project is to make a significant impact on advancing health services research by introducing and testing a novel and potentially powerful service tool that may improve service delivery to address the co-occurring health concerns for women Veterans with any lifetime ST.

DETAILED DESCRIPTION:
The VA Women's Health Research Agenda underscores the importance of improving the safety and health outcomes of returning Veteran women. With greater numbers of women joining the military, the need for gender-specific VA-based interventions is increasingly important. Posttraumatic stress disorder (PTSD), intimate partner violence (IPV), and alcohol use are closely interrelated and significant concerns for women Veterans with a history of sexual trauma (ST). Given that screening for military sexual trauma (MST) is mandated within VAs, a computer delivered intervention has the potential to be easily integrated into the standard of care for women who screen positive for MST and/or other lifetime STs, increasing the identification of high-risk women Veterans. This intervention will provide a computer-based intervention on a VA issued laptop that could improve delivery service and fill a healthcare gap for a vulnerable Veteran population.

The long-term goal of the project is to make a significant impact on advancing health services research by introducing and testing a novel and potentially powerful service tool that may improve service delivery to address the co-occurring health concerns for VA women with lifetime ST. The intervention, Safe and Healthy Experiences (SHE), a brief modular, computer-based intervention, will target interrelated health risks for women Veterans with lifetime ST (i.e. alcohol misuse, IPV, and PTSD). SHE will provide individualized assessment, feedback, and referrals for women Veterans with lifetime ST. The intervention is based on motivational interviewing (MI), a well-defined intervention strategy that has yielded particularly promising results in a range of clinical issues, including interpersonal violence, and a range of patient populations, including male and female Veterans. MI is a collaborative and non-confrontational approach that emphasizes increasing a participant's awareness of successful steps towards well-being. MI is consistent with an empowerment model, which is a highly recommended intervention model for victimized women and both MI and an empowerment model converge on important principles for intervening with victimized women.

Findings from the study will provide the necessary groundwork to examine the efficacy of SHE in a future, large clinical trial. If the SHE intervention is found to be feasible, acceptable and efficacious in improving outcomes for women Veterans with lifetime ST, the ultimate goal would be for the program to be integrated into clinical care and widely disseminated. There are two phases of research directed toward these aims: 1) develop and refine an integrated screening and behavior intervention for VA women with lifetime ST in a brief modular computer-based format that can be administered in a VA primary care setting, and 2) collect data on the feasibility, acceptability, and initial efficacy of the intervention in improving the health of VA women, and increasing utilization of treatment and resources.

The study aims are to:

1. Develop the preliminary computer-based intervention, incorporating information gained in informant interviews.
2. Perform a small open trial (n = 20) of SHE to assess feasibility of recruitment of target population and acceptability of intervention and study procedures.
3. Conduct an initial randomized control trial in a sample of 150 women Veterans who screen positive for lifetime sexual trauma (ST) and have at least one risk factor (i.e., screen positive for intimate partner violence (IPV), posttraumatic stress disorder (PTSD), and/or heavy drinking) to demonstrate the feasibility of SHE and the acceptability of SHE via participant report of ease of use, helpfulness, and overall satisfaction.
4. Examine preliminary evidence for the hypotheses that, relative to the control condition, screening and referral only (SR), SHE will result in:

   * Decreases in the number of risks (i.e., heavy drinking (4+ drinks on one occasion), screen positive for PTSD, screen positive for IPV) at the 2- and 4-month follow-up (primary).
   * Increases in resource and treatment utilization over the 2- and 4-month follow-up period (secondary).

The data will be used to demonstrate whether the effects of the intervention look promising to support a future large-scale randomized control trial and to suggest, in concert with results from clinical trials in related fields, the range of effect sizes that would be reasonable to expect in a future trial.

This is a multi-site study. At the Providence, RI based site (Women and Infants Hospital and Brown University), the specialized computer-based assessment and interactive intervention sessions will be developed and designed and staff members will also assist with data management. The Central Texas VA Healthcare System site will be the data collection site and the main site for participant recruiting, consenting, enrollment, intervention and follow-up. Staff at the two sites will work collaboratively throughout the project to supervise study staff, for reporting to the DOD and IRB's and in designing the assessment and intervention sessions, however, only the study staff at the Central Texas site will have access to participant PHI.

ELIGIBILITY:
Inclusion Criteria:

Female Veterans

* Lifetime history of ST with at least one risk factor: heavy drinking within the past 3 months, screen positive for current PTSD or for IPV within last 12 months
* Age 18-65
* Seeking treatment through the Women's Primary Care Clinics at the Central Texas VA Healthcare System.
* Ability to understand study procedures in English
* Not actively in suicidal or homicidal crisis warranting imminent hospitalization

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2020-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caron Zlotnick, PhD, Principal Investigator — Brown University; Suzannah Creech, PhD, Principal Investigator — VHA VISN 17 COE
Locations (2):
- United States (2):
  - Central Texas Veterans Healthcare System, Temple, Texas
  - Central Texas Veterans Healthcare System, Waco, Texas

IPD SHARING:
Plan to Share IPD: No
No IPD will be made available for sharing

REFERENCES:
- [Derived] O'Doherty L, Whelan M, Carter GJ, Brown K, Tarzia L, Hegarty K, Feder G, Brown SJ. Psychosocial interventions for survivors of rape and sexual assault experienced during adulthood. Cochrane Database Syst Rev. 2023 Oct 5;10(10):CD013456. doi: 10.1002/14651858.CD013456.pub2. PMID 37795783
- [Derived] Creech SK, Pulverman CS, Kahler CW, Orchowski LM, Shea MT, Wernette GT, Zlotnick C. Computerized Intervention in Primary Care for Women Veterans with Sexual Assault Histories and Psychosocial Health Risks: a Randomized Clinical Trial. J Gen Intern Med. 2022 Apr;37(5):1097-1107. doi: 10.1007/s11606-021-06851-0. Epub 2021 May 19. PMID 34013470

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Safety and Health Experiences Program | Control
Started | 76 | 77
Completed | 66 | 69
Not Completed | 10 | 8
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Lost to Follow-up | 10 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Safety and Health Experiences Program | Control | Total
Number analyzed (Participants) | 76 | 77 | 153
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 76 | 77 | 153
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.46 (9.97) | 43.63 (10.28) | 43.55 (10.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 77 | 153
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 12 | 23
  Not Hispanic or Latino | 65 | 65 | 130
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 36 | 37 | 73
  White | 28 | 26 | 54
  More than one race | 2 | 8 | 10
  Unknown or Not Reported | 7 | 5 | 12
Region of Enrollment [Number; unit: participants]
  United States | 76 | 77 | 153

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Health Risks
Description: Number of health risks calculated using scores exceeding threshold on CAS, PCL-5 or AUDIT (see secondary outcomes)
Time Frame: Two months
Population: intent to treat sample
Measure: Mean (Standard Deviation); unit: number of risks
Arm/Group | Safety and Health Experiences Program | Control
Number analyzed (Participants) | 76 | 77
number of risks | 1.38 (.85) | 1.05 (.93)

2. Primary Outcome: Change in Number of Health Risks
Description: Number of health risks calculated using scores exceeding threshold on CAS, PCL-5 or AUDIT (see secondary outcomes)
Time Frame: Four months
Population: intent to treat sample
Measure: Mean (Standard Deviation); unit: number of risks
Arm/Group | Safety and Health Experiences Program | Control
Number analyzed (Participants) | 76 | 77
number of risks | 1.14 (.81) | 1.00 (.81)

3. Secondary Outcome: Adapted Treatment Services Review
Description: Self-report and chart review of utilization of mental health and substance abuse treatment. Range is open, as measure assesses women's self-report of treatment appointments. Higher scores indicate a greater number of treatment appointments and thus greater use of treatment (i.e., better outcome).
Time Frame: 2 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Safety and Health Experiences Program | Control
Number analyzed (Participants) | 76 | 77
score on a scale | 7.32 (10.41) | 3.89 (5.56)

4. Secondary Outcome: Adapted Treatment Services Review
Description: as for outcome 3
Time Frame: 4 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Safety and Health Experiences Program | Control
Number analyzed (Participants) | 76 | 77
score on a scale | 4.59 (7.34) | 5.03 (16.77)

5. Secondary Outcome: The Client Satisfaction Questionnaire
Description: 8-item questionnaire which assesses the participant's satisfaction with the intervention. Score range 4-32; higher scores indicate higher satisfaction with the intervention (i.e., better outcome).
Time Frame: time zero (completed immediately after participant receives intervention session)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- SHE/Safe and Healthy Experiences Intervention: Only women in the intervention group completed the intervention feedback.
Arm/Group | SHE/Safe and Healthy Experiences Intervention
Number analyzed (Participants) | 76
score on a scale | 26.25 (4.0)

6. Other Pre Specified Outcome: Effectiveness in Obtaining Resources Scale
Description: Assesses women's effectiveness in obtaining resources from 11 different types of community resources including church or clergy, health care, legal services, police, or social services. Reporting the subscale for "Things I have been successful at." Score range 0-13; higher scores indicate obtaining more resources (i.e., better outcome).
Time Frame: 2 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Safety and Health Experiences Program | Control
Number analyzed (Participants) | 76 | 77
score on a scale | 1.42 (1.43) | 1.88 (2.17)

7. Other Pre Specified Outcome: Effectiveness in Obtaining Resources Scale
Description: as for outcome 6
Time Frame: 4 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Safety and Health Experiences Program | Control
Number analyzed (Participants) | 76 | 77
score on a scale | 1.48 (1.67) | 1.7 (1.68)

8. Other Pre Specified Outcome: Alcohol Use Disorder Identification Test (AUDIT)
Description: The AUDIT is a 10-item assessment for alcohol use problems, alcohol dependence and problem drinking. Participants respond to each item along 5-point scale ranging from 0 to 4, whereby higher scores reflect more severe alcohol use patterns. Responses are summed to reflect a total score ranging from 0 to 40, with higher scores reflecting higher severity of an individual's use of alcohol.
Time Frame: Four-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Safety and Health Experiences Program | Control
Number analyzed (Participants) | 76 | 77
score on a scale | 4.52 (5.54) | 4.42 (5.01)

9. Other Pre Specified Outcome: Alcohol Use Disorder Identification Test (AUDIT)
Description: as for outcome 8
Time Frame: Two-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Safety and Health Experiences Program | Control
Number analyzed (Participants) | 76 | 77
score on a scale | 4.65 (5.07) | 5.27 (5.60)

10. Other Pre Specified Outcome: Composite Abuse Scale
Description: 30 item measure of chronicity and occurrence of intimate partner violence with current partner in past 12 months. Score range from 0-150; higher scores indicate more intimate partner violence (i.e., worse outcome).
Time Frame: 2 month follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Safety and Health Experiences Program | Control
Number analyzed (Participants) | 45 | 47
score on a scale | 11.25 (13.87) | 6.17 (9.60)

11. Other Pre Specified Outcome: PCL-5
Description: Symptoms of PTSD. Score range 0-80; higher scores indicate more PTSD symptoms (i.e., worse outcome).
Time Frame: 4 month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Safety and Health Experiences Program | Control
Number analyzed (Participants) | 55 | 43
score on a scale | 45.26 (17.01) | 44.81 (18.29)

12. Other Pre Specified Outcome: Composite Abuse Scale
Description: as for outcome 10
Time Frame: 4 month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Safety and Health Experiences Program | Control
Number analyzed (Participants) | 45 | 47
score on a scale | 7.03 (11.76) | 5.48 (10.76)

13. Other Pre Specified Outcome: PCL-5
Description: Symptoms of PTSD. Score range 0-80; higher scores indicate more PTSD symptoms (i.e., worse outcome).
Time Frame: 2 month follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Safety and Health Experiences Program | Control
Number analyzed (Participants) | 55 | 42
score on a scale | 47.16 (17.54) | 42.91 (19.15)

14. Other Pre Specified Outcome: 30-day Alcohol Timeline Follow Back
Description: Calendar-assisted measure used to garner a retrospective account of drinking behavior. Scale is in standard alcoholic drinks in an average week in the past month. Higher numbers indicate more drinks per week (i.e., worse outcome).
Time Frame: 4 month follow-up
Measure: Mean (Standard Deviation); unit: Drinks per week in the past month
Arm/Group | Safety and Health Experiences Program | Control
Number analyzed (Participants) | 28 | 30
Drinks per week in the past month | 8.5 (11.27) | 8.24 (9.03)

15. Other Pre Specified Outcome: 30-day Alcohol Timeline Follow Back
Description: as for outcome 14
Time Frame: 2 month follow up
Measure: Mean (Standard Deviation); unit: Drinks per week in the past month
Arm/Group | Safety and Health Experiences Program | Control
Number analyzed (Participants) | 28 | 30
Drinks per week in the past month | 10.26 (10.84) | 8.26 (9.46)

16. Other Pre Specified Outcome: Satisfaction With CIAS Software Scale
Description: Assesses participant satisfaction with the computerized software with items on likeability, ease of use, level of interest, and respectfulness. Score range is 7-35; higher numbers indicate higher satisfaction with the software (i.e., better outcome).
Time Frame: time zero (completed immediately after participant receives intervention session)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SHE/Safe and Healthy Experiences Intervention
Number analyzed (Participants) | 76
score on a scale | 30.92 (.56)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at 2-month and 4-month follow-up assessments. Timeline of events reported ranges from baseline to 4-month follow-up.
Arm/Group | Safety and Health Experiences Program | Control
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/77
Serious Adverse Events (participants affected / at risk) | 15/76 | 12/77
Other Adverse Events (participants affected / at risk) | 0/76 | 1/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety and Health Experiences Program (N=76) | Control (N=77)
Hospitalization-Vertigo (General disorders) | 0 (0) | 1 (1)
IPV-Physical-Sought no medical care (Injury, poisoning and procedural complications) | 7 (7) | 7 (9)
IPV-Verbal threat (Social circumstances) | 1 (1) | 0 (0)
Hospitalization-Appendicitis (Surgical and medical procedures) | 1 (1) | 0 (0)
Hospitalization-Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Hospitalization-General medical issue (General disorders) | 1 (1) | 2 (2)
Hospitalization-Depression/Heavy drinking (Psychiatric disorders) | 0 (0) | 1 (1)
Hospitalization-Abdominal surgery (Surgical and medical procedures) | 1 (1) | 1 (1)
Hospitalization-General medical issue (Surgical and medical procedures) | 0 (0) | 1 (1)
Sexual assault-Non-IPV (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Physical assault-Non-IPV (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Car accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
IPV-Physical-Doctor's Visit (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hospitalization-Inpatient-Psych (Psychiatric disorders) | 0 (0) | 1 (1)
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety and Health Experiences Program (N=76) | Control (N=77)
Feeling unsafe at home-heard gunshots in neighborhood (Social circumstances) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-26): https://cdn.clinicaltrials.gov/large-docs/47/NCT02957747/Prot_SAP_000.pdf